CLINICAL TRIAL: NCT00616772
Title: Evaluation of Choline Fenofibrate (ABT-335) on Carotid Intima-Media Thickness (cIMT) in Subjects With Type IIb Dyslipidemia With Residual Risk in Addition to Atorvastatin Therapy (FIRST) Trial
Brief Title: Safety and Efficacy Study Using ABT-335 (Investigational Drug) in Combination With Atorvastatin, to Study the Effects on Thickening of the Blood Vessel Wall in Patients With Abnormal Lipid (Fat) Levels in the Blood
Acronym: FIRST
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: AbbVie (prior sponsor, Abbott) (Industry)
Responsible Party: Sponsor
Organization: AbbVie (Industry)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: M10-158
Record Dates: First submitted 2008-02-05; First posted 2008-02-15 (Estimated); Results first posted 2014-01-20 (Estimated); Last update posted 2018-07-02 (Actual); Status verified 2013-12

CONDITIONS: Coronary Artery Disease; Coronary Heart Disease; Dyslipidemia
MeSH Terms: conditions — Coronary Artery Disease; Coronary Disease; Dyslipidemias | interventions — 2-(4-(4-chlorobenzoyl)phenoxy)-2-methylpropanoic acid; fenofibric acid; Atorvastatin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- ABT-335 + Atorvastatin (Experimental): ABT-335 (135 mg) and atorvastatin (up to 40 mg) once daily for 2 years.
  Interventions: Drug: ABT-335; Other: Atorvastatin
- Placebo + Atorvastatin (Placebo Comparator): Placebo and atorvastatin (up to 40 mg) once daily for 2 years.
  Interventions: Drug: Placebo; Other: Atorvastatin

INTERVENTIONS:
Drug: ABT-335 — Capsule
  Other Names: Choline fenofibrate; Fenofibric acid
  Arms: ABT-335 + Atorvastatin
Drug: Placebo — Capsule
  Arms: Placebo + Atorvastatin
Other: Atorvastatin — Capsule

SUMMARY:
The primary purpose of this study is to test the effect and safety of once daily ABT-335 on the thickness of the lining of the carotid artery (a blood vessel to the brain) in patients with abnormal blood lipids who have optimal levels of low density lipoprotein cholesterol ("bad cholesterol") after taking atorvastatin.

ELIGIBILITY:
Inclusion Criteria:

* Patients with mixed dyslipidemia
* Qualifying cIMT thickness

Exclusion Criteria:

* Patients with certain chronic or unstable medical conditions.
* Patients with unstable dose of medications or receiving coumadin, cyclosporine, or certain other medications
* Pregnant or lactating women or women intending to become pregnant
* Patients with diabetes mellitus that is poorly controlled

Min Age: 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 682 (Actual)
Dates: Start 2008-02; Primary Completion 2012-09 (Actual); Study Completion 2012-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Maureen Kelly, MD, Study Director — AbbVie
Locations (124):
- United States (124):
  - Site Reference ID/Investigator# 6747, Chandler, Arizona
  - Site Reference ID/Investigator# 7089, Gilbert, Arizona
  - Site Reference ID/Investigator# 7097, Mesa, Arizona
  - Site Reference ID/Investigator# 26394, Phoenix, Arizona
  - Site Reference ID/Investigator# 6848, Scottsdale, Arizona
  - Site Reference ID/Investigator# 7059, Tempe, Arizona
  - Site Reference ID/Investigator# 7094, Tempe, Arizona
  - Site Reference ID/Investigator# 7098, Tempe, Arizona
  - Site Reference ID/Investigator# 25082, Anaheim, California
  - Site Reference ID/Investigator# 21347, Corona, California
  - Site Reference ID/Investigator# 21483, Garden Grove, California
  - Site Reference ID/Investigator# 21351, Huntington Beach, California
  - Site Reference ID/Investigator# 21346, Laguna Hills, California
  - Site Reference ID/Investigator# 21341, Long Beach, California
  - Site Reference ID/Investigator# 21342, Norwalk, California
  - Site Reference ID/Investigator# 21321, Santa Ana, California
  - Site Reference ID/Investigator# 26242, Tustin, California
  - Site Reference ID/Investigator# 15283, Arvada, Colorado
  - Site Reference ID/Investigator# 7085, Aurora, Colorado
  - Site Reference ID/Investigator# 6749, Denver, Colorado
  - Site Reference ID/Investigator# 7077, Denver, Colorado
  - Site Reference ID/Investigator# 7092, Golden, Colorado
  - Site Reference ID/Investigator# 7722, Littleton, Colorado
  - Site Reference ID/Investigator# 7721, Littleton, Colorado
  - Site Reference ID/Investigator# 11925, Aventura, Florida
  - Site Reference ID/Investigator# 15861, Boynton Beach, Florida
  - Site Reference ID/Investigator# 14422, Deerfield Beach, Florida
  - Site Reference ID/Investigator# 19281, Delray Beach, Florida
  - Site Reference ID/Investigator# 20881, Hollywood, Florida
  - Site Reference ID/Investigator# 20882, Kissimmee, Florida
  - Site Reference ID/Investigator# 19321, Melbourne, Florida
  - Site Reference ID/Investigator# 21353, Melbourne, Florida
  - Site Reference ID/Investigator# 18503, Melbourne, Florida
  - Site Reference ID/Investigator# 18841, Vero Beach, Florida
  - Site Reference ID/Investigator# 19961, Vero Beach, Florida
  - Site Reference ID/Investigator# 7166, West Palm Beach, Florida
  - Site Reference ID/Investigator# 6744, West Palm Beach, Florida
  - Site Reference ID/Investigator# 19301, Atlanta, Georgia
  - Site Reference ID/Investigator# 7051, Atlanta, Georgia
  - Site Reference ID/Investigator# 7109, Atlanta, Georgia
  - Site Reference ID/Investigator# 7326, Dawsonville, Georgia
  - Site Reference ID/Investigator# 7325, Decatur, Georgia
  - Site Reference ID/Investigator# 7057, Dunwoody, Georgia
  - Site Reference ID/Investigator# 7101, Dunwoody, Georgia
  - Site Reference ID/Investigator# 11324, Roswell, Georgia
  - Site Reference ID/Investigator# 6741, Roswell, Georgia
  - Site Reference ID/Investigator# 7103, Suwanee, Georgia
  - Site Reference ID/Investigator# 10761, Addison, Illinois
  - Site Reference ID/Investigator# 6748, Aurora, Illinois
  - Site Reference ID/Investigator# 6742, Aurora, Illinois
  - Site Reference ID/Investigator# 7128, Belleville, Illinois
  - Site Reference ID/Investigator# 7069, Chicago, Illinois
  - Site Reference ID/Investigator# 6849, Chicago, Illinois
  - Site Reference ID/Investigator# 6867, Chicago, Illinois
  - Site Reference ID/Investigator# 6751, Chicago, Illinois
  - Site Reference ID/Investigator# 6847, Chicago, Illinois
  - Site Reference ID/Investigator# 7049, Chicago, Illinois
  - Site Reference ID/Investigator# 7093, Gurnee, Illinois
  - Site Reference ID/Investigator# 6746, Hazel Crest, Illinois
  - Site Reference ID/Investigator# 6743, Melrose Park, Illinois
  - Site Reference ID/Investigator# 7090, Naperville, Illinois
  - Site Reference ID/Investigator# 6750, Oak Brook, Illinois
  - Site Reference ID/Investigator# 6788, Oak Park, Illinois
  - Site Reference ID/Investigator# 6927, Vernon Hills, Illinois
  - Site Reference ID/Investigator# 7076, Erlanger, Kentucky
  - Site Reference ID/Investigator# 8103, Bloomington, Minnesota
  - Site Reference ID/Investigator# 15121, Brooklyn Center, Minnesota
  - Site Reference ID/Investigator# 7050, Edina, Minnesota
  - Site Reference ID/Investigator# 7084, Edina, Minnesota
  - Site Reference ID/Investigator# 6784, City of Saint Peters, Missouri
  - Site Reference ID/Investigator# 6860, St Louis, Missouri
  - Site Reference ID/Investigator# 13182, St Louis, Missouri
  - Site Reference ID/Investigator# 14423, St Louis, Missouri
  - Site Reference ID/Investigator# 14541, St Louis, Missouri
  - Site Reference ID/Investigator# 6740, St Louis, Missouri
  - Site Reference ID/Investigator# 7053, St Louis, Missouri
  - Site Reference ID/Investigator# 7063, Henderson, Nevada
  - Site Reference ID/Investigator# 7070, Henderson, Nevada
  - Site Reference ID/Investigator# 7106, Las Vegas, Nevada
  - Site Reference ID/Investigator# 7518, Las Vegas, Nevada
  - Site Reference ID/Investigator# 7119, Las Vegas, Nevada
  - Site Reference ID/Investigator# 7129, Las Vegas, Nevada
  - Site Reference ID/Investigator# 7071, Cincinnati, Ohio
  - Site Reference ID/Investigator# 7100, Cincinnati, Ohio
  - Site Reference ID/Investigator# 14321, Cincinnati, Ohio
  - Site Reference ID/Investigator# 21355, Cincinnati, Ohio
  - Site Reference ID/Investigator# 7074, Cincinnati, Ohio
  - Site Reference ID/Investigator# 7065, Cincinnati, Ohio
  - Site Reference ID/Investigator# 7075, Dayton, Ohio
  - Site Reference ID/Investigator# 24802, Kettering, Ohio
  - Site Reference ID/Investigator# 7068, Mason, Ohio
  - Site Reference ID/Investigator# 7104, Bellaire, Texas
  - Site Reference ID/Investigator# 7060, Carrollton, Texas
  - Site Reference ID/Investigator# 15282, Dallas, Texas
  - Site Reference ID/Investigator# 6745, Dallas, Texas
  - Site Reference ID/Investigator# 7083, Dallas, Texas
  - Site Reference ID/Investigator# 7127, Dallas, Texas
  - Site Reference ID/Investigator# 7110, Dallas, Texas
  - Site Reference ID/Investigator# 21356, Deer Park, Texas
  - Site Reference ID/Investigator# 11923, Fort Worth, Texas
  - Site Reference ID/Investigator# 7321, Houston, Texas
  - Site Reference ID/Investigator# 21354, Houston, Texas
  - Site Reference ID/Investigator# 21358, Houston, Texas
  - Site Reference ID/Investigator# 26482, Houston, Texas
  - Site Reference ID/Investigator# 7079, Houston, Texas
  - Site Reference ID/Investigator# 7096, Houston, Texas
  - Site Reference ID/Investigator# 7126, Houston, Texas
  - Site Reference ID/Investigator# 8186, Houston, Texas
  - Site Reference ID/Investigator# 11323, Houston, Texas
  - Site Reference ID/Investigator# 7130, Houston, Texas
  - Site Reference ID/Investigator# 11924, Irving, Texas
  - Site Reference ID/Investigator# 13863, Irving, Texas
  - Site Reference ID/Investigator# 7099, McKinney, Texas
  - Site Reference ID/Investigator# 19121, New Braunfels, Texas
  - Site Reference ID/Investigator# 26244, Pearland, Texas
  - Site Reference ID/Investigator# 7105, Plano, Texas
  - Site Reference ID/Investigator# 7061, San Antonio, Texas
  - Site Reference ID/Investigator# 7320, San Antonio, Texas
  - Site Reference ID/Investigator# 7914, San Antonio, Texas
  - Site Reference ID/Investigator# 7058, San Antonio, Texas
  - Site Reference ID/Investigator# 18402, San Antonio, Texas
  - Site Reference ID/Investigator# 7052, San Antonio, Texas
  - Site Reference ID/Investigator# 7062, San Antonio, Texas
  - Site Reference ID/Investigator# 22947, San Antonio, Texas

REFERENCES:
- [Result] Davidson M, Rosenson RS, Maki KC, Nicholls SJ, Ballantyne CM, Setze C, Carlson DM, Stolzenbach J. Study design, rationale, and baseline characteristics: evaluation of fenofibric acid on carotid intima-media thickness in patients with type IIb dyslipidemia with residual risk in addition to atorvastatin therapy (FIRST) trial. Cardiovasc Drugs Ther. 2012 Aug;26(4):349-58. doi: 10.1007/s10557-012-6395-z. PMID 22622962
- See also: Related Info — http://rxabbvie.com

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | ABT-335 + Atorvastatin | Placebo + Atorvastatin
Started | 340 | 342
Treated | 337 | 339
Completed | 225 | 240
Not Completed | 115 | 102

BASELINE CHARACTERISTICS:
Population: All randomized participants who received at least 1 dose of study drug.
Groups:
- Total: Total of all reporting groups
Arm/Group | ABT-335 + Atorvastatin | Placebo + Atorvastatin | Total
Number analyzed (Participants) | 337 | 339 | 676
Age, Continuous [Mean (Standard Deviation); unit: years] | 60.8 (8.71) | 60.7 (8.79) | 60.8 (8.75)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 109 | 109 | 218
  Male | 228 | 230 | 458
Low-density Lipoprotein Cholesterol (LDL-C) [Mean (Standard Deviation); unit: mg/dL] | 84.0 (21.30) | 84.5 (20.47) | 84.3 (20.88)
Triglycerides [Mean (Standard Deviation); unit: mg/dL] | 226.3 (110.01) | 228.7 (127.06) | 227.5 (118.78)
Posterior-wall Carotid Intima-media (cIMT) Thickness [Mean (Standard Deviation); unit: mm] | 0.76 (0.10) | 0.78 (0.12) | 0.77 (0.11)

OUTCOME MEASURES:

1. Primary Outcome: Rate of Change in Mean Posterior-wall Carotid Intima-media Thickness (cIMT)
Description: Rate of change (mm/year) from baseline in mean of posterior-wall carotid intima-media thickness (cIMT) of the left and right common carotid artery. The statistical model used change from baseline as the dependent variable, with time of cIMT assessment (in years) as one of the factors in the model. The between-group difference in the rate of change was based on the parameter coefficient for the time-by-treatment interaction. The within-group rate of change was obtained from estimate statements within the repeated measures analysis. cIMT was measured using non-invasive ultrasound.
Time Frame: Baseline, 6 months, 12 months, 18 months, and 24 months
Population: All randomized participants who had both a baseline value and at least 1 postbaseline value for that parameter.
Measure: Mean (Standard Error); unit: mm/year
Arm/Group | ABT-335 + Atorvastatin | Placebo + Atorvastatin
Number analyzed (Participants) | 281 | 291
mm/year | -0.006 (0.0037) | 0.000 (0.0036)
Statistical Analysis 1: Comparison: ABT-335 + Atorvastatin vs Placebo + Atorvastatin; Test type: Superiority or Other; p = 0.220, Repeated measures linear mixed model; Fixed effects for baseline cIMT, baseline atorvastatin dose, central imaging site, treatment group, time; interaction between treatment group and time; Mean Difference (Final Values) = -0.006, 95% CI 2-sided [-0.016 to 0.004]

2. Secondary Outcome: Rate of Change in Mean of Maximal Posterior-wall Carotid Intima-media Thickness (cIMT)
Description: Rate of change (mm/year) from baseline in mean of maximal posterior-wall carotid intima-media thickness (cIMT) of the left and right common carotid artery. The statistical model used change from baseline as the dependent variable, with time of cIMT assessment (in years) as one of the factors in the model. The between-group difference in the rate of change was based on the parameter coefficient for the time-by-treatment interaction. The within-group rate of change was obtained from estimate statements within the repeated measures analysis. cIMT was measured using non-invasive ultrasound.
Time Frame: Baseline, 6 months, 12 months, 18 months, and 24 months
Population: All randomized subjects who had both a baseline value and at least 1 postbaseline value for that parameter.
Measure: Mean (Standard Error); unit: mm/year
Arm/Group | ABT-335 + Atorvastatin | Placebo + Atorvastatin
Number analyzed (Participants) | 281 | 291
mm/year | -0.005 (0.0047) | -0.003 (0.0046)
Statistical Analysis 1: Comparison: ABT-335 + Atorvastatin vs Placebo + Atorvastatin; Test type: Superiority or Other; p = 0.813, Repeated measures linear mixed model; Fixed effects for baseline atorvastatin dose, imaging site, treatment, time; interaction between treatment group and time; baseline cIMT as covariate; Mean Difference (Final Values) = -0.002, 95% CI 2-sided [-0.014 to 0.011]

3. Secondary Outcome: Rate of Change in Composite of Mean of the Mean Posterior-wall Intima-media Thickness (IMT)
Description: Rate of change (mm/year) from baseline in composite of mean of the mean posterior-wall intima-media thickness (IMT) of the left and right common carotid artery, internal carotid artery, and carotid bifurcation. The statistical model used change from baseline as the dependent variable, with time of IMT assessment (in years) as one of the factors in the model. The between-group difference in the rate of change was based on the parameter coefficient for the time-by-treatment interaction. The within-group rate of change was obtained from estimate statements within the repeated measures analysis. IMT was measured using non-invasive ultrasound.
Time Frame: Baseline, 6 months, 12 months, 18 months, and 24 months
Population: All randomized subjects who had both a baseline value and at least 1 postbaseline value for that parameter, as well as 3 or more matching segments at baseline and the 2-year visit. Observations at the interim visits were included only if 3 or more segments matched the segments at baseline and at 2 years.
Measure: Mean (Standard Error); unit: mm/year
Arm/Group | ABT-335 + Atorvastatin | Placebo + Atorvastatin
Number analyzed (Participants) | 138 | 133
mm/year | -0.010 (0.0039) | -0.004 (0.0041)
Statistical Analysis 1: Comparison: ABT-335 + Atorvastatin vs Placebo + Atorvastatin; Test type: Superiority or Other; p = 0.249, Repeated measures linear mixed model; Fixed effects for baseline atorvastatin dose, imaging site, treatment, time; interaction between treatment group and time; baseline IMT as covariate; Mean Difference (Final Values) = -0.007, 95% CI 2-sided [-0.018 to 0.005]

4. Secondary Outcome: Rate of Change in Composite of Mean of Maximal Posterior-wall Intima-media Thickness (IMT)
Description: Rate of change (mm/year) from baseline in composite of mean of maximal posterior-wall intima-media thickness (IMT) of the left and right common carotid artery, internal carotid artery, and carotid bifurcation. The statistical model used change from baseline as the dependent variable, with time of IMT assessment (in years) as one of the factors in the model. The between-group difference in the rate of change was based on the parameter coefficient for the time-by-treatment interaction. The within-group rate of change was obtained from estimate statements within the repeated measures analysis. IMT was measured using non-invasive ultrasound.
Time Frame: Baseline, 6 months, 12 months, 18 months, and 24 months
Population: as for outcome 3
Measure: Mean (Standard Error); unit: mm/year
Arm/Group | ABT-335 + Atorvastatin | Placebo + Atorvastatin
Number analyzed (Participants) | 138 | 133
mm/year | -0.014 (0.0053) | -0.008 (0.0056)
Statistical Analysis 1: Comparison: ABT-335 + Atorvastatin vs Placebo + Atorvastatin; Test type: Superiority or Other; p = 0.487, Repeated measures linear mixed model; [statistical method as in outcome 3, analysis 1]; Mean Difference (Final Values) = -0.005, 95% CI 2-sided [-0.020 to 0.010]

5. Secondary Outcome: Rate of Change in Composite of Mean of Maximal Posterior-wall and Anterior-wall Intima-media Thickness (IMT)
Description: Rate of change (mm/year) from baseline in composite of mean of maximal posterior-wall and anterior-wall intima-media thickness (IMT) of the left and right common carotid artery, internal carotid artery, and carotid bifurcation. The statistical model used change from baseline as the dependent variable, with time of IMT assessment (in years) as one of the factors in the model. The between-group difference in the rate of change was based on the parameter coefficient for the time-by-treatment interaction. The within-group rate of change was obtained from estimate statements within the repeated measures analysis. IMT was measured using non-invasive ultrasound.
Time Frame: Baseline, 6 months, 12 months, 18 months, and 24 months
Population: All randomized subjects who had both a baseline value and at least 1 postbaseline value for that parameter, as well as 6 or more matching segments at baseline and the 2-year visit. Observations at the interim visits were included only if 6 or more segments matched the segments at baseline and at 2 years.
Measure: Mean (Standard Error); unit: mm/year
Arm/Group | ABT-335 + Atorvastatin | Placebo + Atorvastatin
Number analyzed (Participants) | 67 | 66
mm/year | -0.003 (0.0070) | -0.019 (0.0067)
Statistical Analysis 1: Comparison: ABT-335 + Atorvastatin vs Placebo + Atorvastatin; Test type: Superiority or Other; p = 0.112, Repeated measures linear mixed model; [statistical method as in outcome 3, analysis 1]; Mean Difference (Final Values) = 0.016, 95% CI 2-sided [-0.004 to 0.035]

ADVERSE EVENTS:
Time Frame: AEs that occurred on or after the first dose of study drug through 30 days after last dose of study drug (up to 25 months).
Arm/Group | ABT-335 + Atorvastatin | Placebo + Atorvastatin
Serious Adverse Events (participants affected / at risk) | 58/337 | 66/339
Other Adverse Events (participants affected / at risk) | 235/337 | 241/339
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | ABT-335 + Atorvastatin (N=337) | Placebo + Atorvastatin (N=339)
COAGULOPATHY (Blood and lymphatic system disorders) | 1 | 0
ACUTE CORONARY SYNDROME (Cardiac disorders) | 1 | 0
ACUTE MYOCARDIAL INFARCTION (Cardiac disorders) | 2 | 1
ANGINA PECTORIS (Cardiac disorders) | 0 | 1
ANGINA UNSTABLE (Cardiac disorders) | 1 | 0
ATRIAL FIBRILLATION (Cardiac disorders) | 0 | 1
ATRIOVENTRICULAR BLOCK COMPLETE (Cardiac disorders) | 1 | 1
CARDIAC FAILURE (Cardiac disorders) | 0 | 1
CARDIAC FAILURE CONGESTIVE (Cardiac disorders) | 2 | 1
CORONARY ARTERY DISEASE (Cardiac disorders) | 6 | 5
CORONARY ARTERY STENOSIS (Cardiac disorders) | 0 | 2
DIASTOLIC DYSFUNCTION (Cardiac disorders) | 0 | 1
EXTRASYSTOLES (Cardiac disorders) | 1 | 0
ISCHAEMIC CARDIOMYOPATHY (Cardiac disorders) | 0 | 1
MYOCARDIAL INFARCTION (Cardiac disorders) | 3 | 1
MYOCARDIAL ISCHAEMIA (Cardiac disorders) | 0 | 1
PERICARDITIS (Cardiac disorders) | 0 | 1
SUPRAVENTRICULAR TACHYCARDIA (Cardiac disorders) | 1 | 0
TACHYARRHYTHMIA (Cardiac disorders) | 1 | 0
VENTRICULAR TACHYCARDIA (Cardiac disorders) | 1 | 0
WOLFF-PARKINSON-WHITE SYNDROME (Cardiac disorders) | 0 | 1
VERTIGO (Ear and labyrinth disorders) | 2 | 1
VESTIBULAR DISORDER (Ear and labyrinth disorders) | 1 | 0
RETINAL HAEMORRHAGE (Eye disorders) | 0 | 1
ABDOMINAL HERNIA (Gastrointestinal disorders) | 0 | 1
COLITIS ISCHAEMIC (Gastrointestinal disorders) | 1 | 0
DIARRHOEA (Gastrointestinal disorders) | 1 | 0
DIVERTICULUM INTESTINAL HAEMORRHAGIC (Gastrointestinal disorders) | 1 | 0
GASTROINTESTINAL HAEMORRHAGE (Gastrointestinal disorders) | 1 | 1
GASTROOESOPHAGEAL REFLUX DISEASE (Gastrointestinal disorders) | 1 | 1
INGUINAL HERNIA (Gastrointestinal disorders) | 1 | 0
LOWER GASTROINTESTINAL HAEMORRHAGE (Gastrointestinal disorders) | 0 | 1
NAUSEA (Gastrointestinal disorders) | 1 | 0
PANCREATITIS ACUTE (Gastrointestinal disorders) | 1 | 0
SMALL INTESTINAL OBSTRUCTION (Gastrointestinal disorders) | 1 | 0
VOMITING (Gastrointestinal disorders) | 1 | 0
CHEST PAIN (General disorders) | 1 | 1
MEDICAL DEVICE COMPLICATION (General disorders) | 1 | 0
NON-CARDIAC CHEST PAIN (General disorders) | 4 | 3
CHOLECYSTITIS (Hepatobiliary disorders) | 1 | 1
CHOLECYSTITIS ACUTE (Hepatobiliary disorders) | 1 | 0
CHOLELITHIASIS (Hepatobiliary disorders) | 0 | 1
ABSCESS (Infections and infestations) | 0 | 1
ARTHRITIS INFECTIVE (Infections and infestations) | 1 | 0
BRONCHITIS (Infections and infestations) | 0 | 1
CELLULITIS (Infections and infestations) | 1 | 0
CLOSTRIDIAL INFECTION (Infections and infestations) | 1 | 0
DIVERTICULITIS (Infections and infestations) | 2 | 0
PNEUMONIA (Infections and infestations) | 4 | 3
PYELONEPHRITIS (Infections and infestations) | 1 | 0
SIALOADENITIS (Infections and infestations) | 1 | 0
STAPHYLOCOCCAL INFECTION (Infections and infestations) | 0 | 1
STAPHYLOCOCCAL SEPSIS (Infections and infestations) | 0 | 1
ANKLE FRACTURE (Injury, poisoning and procedural complications) | 2 | 2
FOOT FRACTURE (Injury, poisoning and procedural complications) | 1 | 0
HEAD INJURY (Injury, poisoning and procedural complications) | 0 | 1
HUMERUS FRACTURE (Injury, poisoning and procedural complications) | 0 | 1
JAW FRACTURE (Injury, poisoning and procedural complications) | 0 | 1
MENISCUS LESION (Injury, poisoning and procedural complications) | 0 | 1
MULTIPLE INJURIES (Injury, poisoning and procedural complications) | 1 | 0
MUSCLE RUPTURE (Injury, poisoning and procedural complications) | 0 | 1
ROAD TRAFFIC ACCIDENT (Injury, poisoning and procedural complications) | 2 | 0
UPPER LIMB FRACTURE (Injury, poisoning and procedural complications) | 0 | 1
BLOOD CREATINE PHOSPHOKINASE INCREASED (Investigations) | 1 | 0
BLOOD CREATININE INCREASED (Investigations) | 0 | 1
DEHYDRATION (Metabolism and nutrition disorders) | 1 | 0
HYPERGLYCAEMIA (Metabolism and nutrition disorders) | 1 | 1
ARTHRALGIA (Musculoskeletal and connective tissue disorders) | 3 | 2
ARTHRITIS (Musculoskeletal and connective tissue disorders) | 1 | 0
CERVICAL SPINAL STENOSIS (Musculoskeletal and connective tissue disorders) | 0 | 1
INTERVERTEBRAL DISC PROTRUSION (Musculoskeletal and connective tissue disorders) | 0 | 1
JOINT INSTABILITY (Musculoskeletal and connective tissue disorders) | 1 | 0
MUSCULOSKELETAL CHEST PAIN (Musculoskeletal and connective tissue disorders) | 0 | 1
OSTEOARTHRITIS (Musculoskeletal and connective tissue disorders) | 2 | 1
BENIGN PANCREATIC NEOPLASM (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
BRAIN NEOPLASM BENIGN (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
BREAST CANCER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
BREAST CANCER IN SITU (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
CARCINOID TUMOUR PULMONARY (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
ENDOMETRIAL CANCER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
LARGE CELL CARCINOMA OF THE RESPIRATORY TRACT STAGE UNSPECIFIED (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
METASTATIC NEOPLASM (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
NEUROENDOCRINE CARCINOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
NON-SMALL CELL LUNG CANCER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
OESOPHAGEAL CARCINOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
OVARIAN CANCER STAGE III (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
PROSTATE CANCER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 1
PROSTATE CANCER STAGE II (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
SARCOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
CEREBROVASCULAR ACCIDENT (Nervous system disorders) | 0 | 2
CERVICOBRACHIAL SYNDROME (Nervous system disorders) | 0 | 1
COMPLICATED MIGRAINE (Nervous system disorders) | 1 | 0
DIABETIC NEUROPATHY (Nervous system disorders) | 1 | 0
ISCHAEMIC STROKE (Nervous system disorders) | 0 | 1
METABOLIC ENCEPHALOPATHY (Nervous system disorders) | 1 | 0
PRESYNCOPE (Nervous system disorders) | 1 | 0
RUPTURED CEREBRAL ANEURYSM (Nervous system disorders) | 1 | 0
SYNCOPE (Nervous system disorders) | 1 | 3
TRANSIENT ISCHAEMIC ATTACK (Nervous system disorders) | 1 | 3
UNRESPONSIVE TO STIMULI (Nervous system disorders) | 0 | 1
GENERALISED ANXIETY DISORDER (Psychiatric disorders) | 0 | 1
MAJOR DEPRESSION (Psychiatric disorders) | 1 | 1
SUICIDAL IDEATION (Psychiatric disorders) | 1 | 0
NEPHROLITHIASIS (Renal and urinary disorders) | 0 | 1
NEPHROTIC SYNDROME (Renal and urinary disorders) | 0 | 1
RENAL FAILURE ACUTE (Renal and urinary disorders) | 3 | 0
BENIGN PROSTATIC HYPERPLASIA (Reproductive system and breast disorders) | 0 | 1
ACUTE RESPIRATORY FAILURE (Respiratory, thoracic and mediastinal disorders) | 1 | 0
ASTHMA (Respiratory, thoracic and mediastinal disorders) | 0 | 1
CHRONIC OBSTRUCTIVE PULMONARY DISEASE (Respiratory, thoracic and mediastinal disorders) | 2 | 1
HYPOXIA (Respiratory, thoracic and mediastinal disorders) | 0 | 1
NASAL POLYPS (Respiratory, thoracic and mediastinal disorders) | 0 | 1
PULMONARY EMBOLISM (Respiratory, thoracic and mediastinal disorders) | 1 | 1
PULMONARY MASS (Respiratory, thoracic and mediastinal disorders) | 1 | 1
RESPIRATORY FAILURE (Respiratory, thoracic and mediastinal disorders) | 1 | 1
ANGIOEDEMA (Skin and subcutaneous tissue disorders) | 0 | 1
ANEURYSM (Vascular disorders) | 1 | 0
AORTIC ANEURYSM (Vascular disorders) | 1 | 2
AORTIC STENOSIS (Vascular disorders) | 1 | 1
FEMORAL ARTERY OCCLUSION (Vascular disorders) | 1 | 0
PERIPHERAL ARTERIAL OCCLUSIVE DISEASE (Vascular disorders) | 0 | 2
PERIPHERAL VASCULAR DISORDER (Vascular disorders) | 1 | 1
SUBCLAVIAN ARTERY ANEURYSM (Vascular disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | ABT-335 + Atorvastatin (N=337) | Placebo + Atorvastatin (N=339)
CONSTIPATION (Gastrointestinal disorders) | 17 | 14
DIARRHOEA (Gastrointestinal disorders) | 23 | 25
NAUSEA (Gastrointestinal disorders) | 24 | 20
FATIGUE (General disorders) | 23 | 17
OEDEMA PERIPHERAL (General disorders) | 15 | 19
BRONCHITIS (Infections and infestations) | 24 | 30
NASOPHARYNGITIS (Infections and infestations) | 44 | 38
SINUSITIS (Infections and infestations) | 20 | 30
UPPER RESPIRATORY TRACT INFECTION (Infections and infestations) | 53 | 58
URINARY TRACT INFECTION (Infections and infestations) | 18 | 14
BLOOD CREATININE INCREASED (Investigations) | 22 | 6
DIABETES MELLITUS (Metabolism and nutrition disorders) | 27 | 11
ARTHRALGIA (Musculoskeletal and connective tissue disorders) | 29 | 36
BACK PAIN (Musculoskeletal and connective tissue disorders) | 36 | 43
MUSCLE SPASMS (Musculoskeletal and connective tissue disorders) | 24 | 23
MUSCULOSKELETAL PAIN (Musculoskeletal and connective tissue disorders) | 22 | 15
MYALGIA (Musculoskeletal and connective tissue disorders) | 26 | 32
PAIN IN EXTREMITY (Musculoskeletal and connective tissue disorders) | 44 | 26
DIZZINESS (Nervous system disorders) | 29 | 20
HEADACHE (Nervous system disorders) | 38 | 43
INSOMNIA (Psychiatric disorders) | 18 | 20
COUGH (Respiratory, thoracic and mediastinal disorders) | 23 | 18
HYPERTENSION (Vascular disorders) | 17 | 36

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
AbbVie requests that any investigator or institution that plans on presenting/publishing results disclosure, provide written notification of their request 60 days prior to their presentation/publication. AbbVie requests that no presentation/publication will be instituted until 12 months after a study is completed, or after the first presentation/publication whichever occurs first. A delay may be proposed of a presentation/publication if AbbVie needs to secure patent or proprietary protection.